CLINICAL TRIAL: NCT03528057
Title: Randomized, Prospective Evaluation of Hemostatic Agents in Robotic-assisted Laparoscopic Partial Nephrectomy
Brief Title: Evaluation of Hemostatic Agents in Robotic-assisted Laparoscopic Partial Nephrectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting participants.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert B. Nadler, Vice Chair, Department of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00206993
Record Dates: First submitted 2018-04-18; First posted 2018-05-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Robotic-Assisted Laparoscopic Partial Nephrectomy; Hemostatic Agents; Renal Malignant Tumor
Keywords: Kidney
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgical team and the patient will be blinded as to which arm the patient will be assigned both at the time of recruitment in the clinic and at the start of surgery. The patient and surgeon will both be blinded at the start of the surgery (RALPN). The surgeon will be informed intra-operatively during the renorrhaphy portion of the procedure as to which arm the patient will be assigned, at which point he will be un-blinded. Following completion of the entire surgery, the patient will also be informed as to which arm he/she was randomized upon request.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (Active Comparator): Patients undergoing RALPN with the use of HAs by a surgeon.
  Interventions: Device: Hemostat
- Group 2 (No Intervention): Patients undergoing RALPN without the use of HAs by a surgeon

INTERVENTIONS:
Device: Hemostat — Hemostatic agents, if used at all during surgery, will be applied laparoscopically into the tumor bed to stop bleeding. The type of hemostat will be decided by the surgeon according to the anatomy of the tumor bed.
  Other Names: Surgicel Nu-Knit; FLOSEAL Hemostatic Matrix
  Arms: Group 1

SUMMARY:
The aim of this study is to evaluate whether Hemostatic Agents (HA) make a significant clinical difference in patient outcomes when used for Robotic-Assisted Laparoscopic Partial Nephrectomy (RALPN). The result of this trial will determine whether HAs are necessary for use during RALPN or if they can be omitted from the surgical tools available during this procedure. This study has a direct clinical implication on a patient's outcomes following RALPN, specifically whether patients will have better, worse, or unchanged outcomes with RALPN if HAs are used.

DETAILED DESCRIPTION:
Partial nephrectomy is a surgical procedure wherein a diseased segment of a kidney is surgically removed, leaving behind the remaining healthy kidney parenchyma. This surgical procedure is typically performed to remove mass lesions suspicious for malignancy. A major goal of partial nephrectomy is to spare as much renal function as possible by preserving the healthy portion of the kidney while removing only the pathologic portion of the kidney.

Hemostatic agents (HA) are devices commonly used during robotic-assisted laparoscopic partial nephrectomy (RALPN) due to the risk of bleeding posed by incising a highly vascular organ. The use of various HAs as part of the surgical technique for RALPN is well-described. Potential benefits such as lower blood loss, lower rate of urine leak, and lower blood product transfusion rates have been suggested in small case series. However, larger prospective studies have failed to demonstrate these benefits of HAs. They report similar patient outcomes regardless of HA use. However, these studies are subject to selection bias given the lack of randomization, and they had a small relative number of partial nephrectomies performed without HAs.

To the knowledge of the investigators, no randomized trials have addressed the use of HAs in RALPN. Randomized, controlled trials for partial hepatectomy and knee arthroplasty have shown no benefit when using hemostatic agents to control bleeding.

At the home institution for this study, surgeons routinely use HAs in the resection bed during RALPN. Available, FDA approved, commercial agents include Floseal and Nu-Knit®. Each unit of HA costs $150 - $419 per unit, and often multiple units are used during a given procedure. The hospital is paid a set amount based on the patient's insurance for performing the procedure regardless of use of HA. The use of HAs therefore increases costs incurred by the hospital when performing these procedures. It is imperative to determine if this expenditure is justified.

The primary aim of this study is to compare surgical outcomes in patients undergoing RALPN with and without the use of hemostatic agents. Given the small nature of and conflicting information from the aforementioned cohort studies, it is imperative to remove selection bias and perform a randomized comparison of HA use. This study will provide a much more definitive head-to-head comparison of the overall utility of HAs. Additionally, it may provide more information about differential patient selection for more appropriate and judicious use of HAs. No study has evaluated differential patient selection for HA use, and therefore any finding in this realm would be novel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older.
* Patients must have a solid or cystic renal mass suspicious for malignancy by imaging with ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI).
* Patients must be initially scheduled RALPN as opposed to radical nephrectomy or other techniques for partial nephrectomy such as open surgery or pure laparoscopy without robot assistance.
* Patients with bilateral kidneys or a solitary kidney, so long as these are native kidneys as opposed to a transplanted kidney.
* Patients can have the common single renal artery and single renal vein, or they can have common variants such as two renal arteries and/or two renal veins.

Exclusion Criteria:

* Patients on hemodialysis.
* Patients who have had a renal transplantation.
* Patients on therapeutic anticoagulation prior to surgery (example anticoagulants include: aspirin 325 mg daily, clopidogrel, warfarin, fondaparinux, dabigatran, and rivaroxaban). However, patients who take aspirin 81 mg daily as their daily regimen will be included.
* Patients with bleeding disorders (example: hemophilia) and other documented coagulopathy (example: chronic liver disease) with international normalized ratio (INR) > 1.0 at baseline.
* Patients who have had a prior surgical procedure, aside from percutaneous renal biopsy, on the kidney in the current operation.
* Patients with over 100 mL of estimated blood loss (calculated by anesthesia team using the suction canisters) prior to clamping of the renal hilum will be excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Absolute change in hemoglobin | Morning after surgery
  This will be measured as the difference between the hemoglobin obtained postoperatively (measured at approximately 4 am in the morning after surgery) and the hemoglobin obtained preoperatively in the holding area on the day of surgery.

SECONDARY OUTCOMES:
Total number of major bleeding complications | 30 days following surgery
  Major complications are blood loss requiring transfusion of packed red blood cells, reoperation, and endovascular ablation
Safety monitoring parameters | 30 days following surgery
  Incidence of any of the following: urine leak, stroke, cardiac arrest, myocardial infarction, and death.
Operating room parameters | Total duration of surgery
  The number of sutures used during renorrhaphy and capsular closure.
Operating room parameters | Total duration of surgery
  Duration of renorrhaphy.
Operating room parameters | Total duration of surgery
  Number of patients in Group 2 (no HA) who required HA at the surgeon's discretion.
Total length of in-patient hospital stay | 30 days following surgery
  Total length of all inpatient hospital stay over 30 days measured in days.
Total charges | 30 days following surgery
  Total charges for all inpatient care over 30 days using billing information recorded in the Northwestern Electronic Data Warehouse.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nadler, MD, Principal Investigator — Professor of Urology, Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States